CLINICAL TRIAL: NCT02095496
Title: Contribution to the Understanding of the Involvement of Mechanical Ventilation in ICU Patients Sleep Disorders
Brief Title: Efficacy of Closed-loop Ventilation to Reduced Sleep Disorders
Acronym: SleepICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: StLuc
Record Dates: First submitted 2014-03-04; First posted 2014-03-24 (Estimated); Last update posted 2016-02-01 (Estimated); Status verified 2016-01

CONDITIONS: Acute Mechanical Ventilatory Failure; Psychosis Associated With Intensive Care
Keywords: sleep; intensive care; mechanical ventilation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intellivent-ASV (Experimental): Patients will receive Intellivent-ASV ventilation during 12 hours
  Interventions: Device: Intellivent-ASV
- Conventional ventilation (Active Comparator): Patients will receive pressure support ventilation during 12 hours
  Interventions: Device: Conventional ventilation

INTERVENTIONS:
Device: Intellivent-ASV — 12 hours of mechanical ventilation with intellivent-ASV
  Other Names: closed-loop ventilation
  Arms: Intellivent-ASV
Device: Conventional ventilation — 12 hours of mechanical ventilation with pressure support ventilation
  Other Names: pressure support ventilation
  Arms: Conventional ventilation

SUMMARY:
Sleep's deficiencies are very common in intensive care. Mechanical ventilation is a known factor in this deterioration.The investigators hypothesize that close-loop ventilation mode (Intellivent-ASV) is able to minimize sleep deterioration, adjusting ventilation to the patient needs.

DETAILED DESCRIPTION:
In intensive care, conventional mechanical ventilation (pressure support) generates apneas and asynchronies during sleep. Intellivent-ASV would be able to avoid apneas, providing controlled cycles when respiratory rate become too low. Moreover, the constant adjustment of ventilatory parameters to the patient needs would avoid asynchronies between the ventilator and the patient ventilatory drive.

ELIGIBILITY:
Inclusion Criteria:

* patient under invasive mechanical ventilation since at least 6 hours and for expected at least 48 hours duration, including a continuous period of 24h, from 2 p.m. to 2 p.m. the next day.
* Age > 18 years
* Body Mass Index < 40
* informed consent signed by the family

Exclusion Criteria:

* patient requiring neuo-muscular blocking agent or deep sedation enough to abolish spontaneous ventilatory effort
* patient with encephalopathy regardless of origin
* Patient with Glasgow coma scale score < 8
* Patient abusing of drug or alcohol
* patient with a contraindication for placement of a nasogastric tube such that sufferers of esophageal or gastric ulcer, tumors, diverticulitis or bleeding varices or patients with sinusitis epistaxis or having recently been operated on the nose or pharynx
* Patient with bleeding disorders
* Patient with unstable respiratory situation as defined by a arterial oxygen partial pressure and inspired oxygen fraction ratio (PaO2/FiO2) < 100 mmHg with positive end expiratory pressure (PEEP) > 12 cmH2O
* Patient with unstable hemodynamic situation as defined by Systolic Blood Pressure (SBP) < 75 mmHg despite a therapeutic optimization
* Inclusion in another research protocol submitted to consent

Ages: 18 Years to 94 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Sleep fragmentation index | 12 hours
  = number of awakenings and arousals per hour of sleep

SECONDARY OUTCOMES:
duration of sleep episodes | 12 hours
Distribution of the sleep | 12 hours
  distribution of the sleep during day and night

OTHER OUTCOMES:
Sleep's architecture | 12 hours
  proportion of the different phases of sleep (slow waves sleep stage 1, 2, 3 and 4 and Rapid Eye Movement (REM) sleep)
ventilation | 12 hours
  number of asynchronies and apneas and ventilatory variability
circadian rhythm | 6 hours
  Plasmatic melatonin dosage

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Bialais, PhD Student, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Intensive Care Unit, Saint Luc university Hospital, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No